CLINICAL TRIAL: NCT06505018
Title: A Randomized Phase III Study Comparing the Digital Telemonitoring Platform "CUREETY TECHCARE" to Usual Standard of Care in Patients With Triple Negative Metastatic Breast Cancer Initiating a First-line Systemic Treatment
Brief Title: Telemonitoring Platform "CUREETY TECHCARE" vs Standard of Care for mTBNC Patients Initiating a First-line Treatment
Acronym: ALTERNATIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Cureety (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UC-BCG-2309; IDRCB NUMBER: 2023-A02477-38 (Other: CPP Sud-Méditerranée III)
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Triple-Negative Breast Carcinoma
Keywords: Telemonitoring; Triple Negative Breast Cancer; Cureety; Adverse events
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring group (Experimental): Standard of care with digital telemonitoring "Cureety TechCare". The telemonitoring will comprise weekly adverse event (AE) evaluations and their analyses by the "Cureety TechCare".
  Interventions: Device: Cureety techcare
- Standard-of-care group (No Intervention)

INTERVENTIONS:
Device: Cureety techcare — Each week, patients complete a questionnaire via the Cureety platform, specifically designed for the drug class or specific treatment being administered. Based on their responses, the Cureety TechCare algorithm classifies patients into one of four risk categories: "correct" (green), "compromised" (yellow), "state to be monitored" (orange), or "critical state" (red). (Note: the color code is not visible to the patient).
  The medical team uses the dashboard for daily patient monitoring and manages alerts related to the "clinical classification" of the patient's condition. The physician in charge of telemonitoring interprets the data, adjusts the treatment as needed, and provides supportive care during standard care consultations. Patients are also notified of alerts with tailored messages guiding them on the actions to take according to the category determined by the device.
  Arms: Telemonitoring group

SUMMARY:
The goal of this clinical trial is to assess whether adding telemonitoring (the digital telemonitoring platform "CUREETY TECHCARE"), to standard care, will benefit patients with previously untreated metastatic triple-negative breast cancer starting first-line cancer therapy.

The main questions it aims to answer are:

* Is patient quality of life improved by using the telemonitoring platform?
* Are patients hospitalized less frequently when using the telemonitoring platform?
* Is the patient overall survival improved by telemonitoring ?

Researchers will compare data from patients using telemonitoring while receiving standard care with data from patients receiving only standard care.

Participants using telemonitoring will answer questions about their symptoms on the platform. The platform will analyze these symptoms, assess the patient's general condition and provide advice accordingly. Medical staff will also access the platform to monitor the patient's general condition and contact them if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Signed a written informed consent form prior to participate in the study. Note: In case of physical incapacitation, a trusted representative of their choice, which is not the Investigator or sponsor, can sign on the behalf of the patients
* Patients ≥18 years of age.
* Patient with histologically documented metastatic triple negative breast cancer (ER (Oestrogen receptor) and PR (Progesterone receptor) <10%, Her2 negative status).
* Life expectancy > 6 months as per investigator estimate.
* Patient initiating a marketed authorized first-line systemic treatment in the metastatic setting.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2.
* Patient having completed the EORTC QLQ-C30 and EORTC QLQ-BR45 at baseline (response to questions 29 and 30 of EORTC QLQ-C30 at baseline are mandatory)
* Affiliated to the social security system or equivalent health insurance.
* Patient able and willing to complete web-based self-reported questionnaires, from initiation of first-line treatment and for the duration of the study (over multiple treatment lines)
* Patient has access to a computer, tablet, or smartphone connected to the Internet.

Exclusion Criteria:

* Participation in another clinical trial using telemonitoring.
* Physical or psychological incapacity of the patient to use the digital telemonitoring Cureety Techcare, according to the investigator's discretion.
* Patient deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-02 (Estimated)

PRIMARY OUTCOMES:
Time to definitive Health-Related Quality of life score Deterioration | At baseline then every 3 months, up to 24 months
  The time to definitive Health-Related Quality of life score Deterioration is the length of time from randomization to the first deterioration of ≥ 10 points out of 100 or ≥2 points out of 14 in the global health status (GHS) score (items 29 and 30 of the QLQ-C30) compared with the baseline, assuming no improvement of at least 2 points in the GHS score compared with the baseline has occurred.
  The responses to the items 29-30 of the QLQ-C30 will be scored using the QLQ scoring manual. These 2 items have possible values ranging from 1 (very bad) to 7 (excellent) corresponding to a sum from 2 to 14 points. After conversion to percentages, the GHS will range from 0% to 100%. The higher the value, the better the quality of life.
Hospitalization-free survival | From randomization to death from any cause, up to 24 months
  Hospitalization-free survival is the length of time from randomization during which patients enrolled in the study are not hospitalized and remain alive.
Overall survival | From randomization to death from any cause, up to 24 months after last inclusion
  overall survival is the length of time from randomization during which patients enrolled in the study remain alive.

SECONDARY OUTCOMES:
Time-to-treatment failure | From randomization to treatment discontinuation, up to 24 months
  Time-to-treatment failure is the time interval (in months) between the initiation of first-line chemotherapy and its premature discontinuation, irrespective of the reason for discontinuation.
Toxicity-free survival | From randomization until the first event, up to 24 months
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the oncology research community as the leading rating scale for adverse events. This scale, divided into five grades (1 = "mild," 2 = "moderate," 3 = "severe," 4 = "life-threatening," and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders. Toxicity-free survival is defined as the time from randomization to the first event among a grade 3-4 non-hematological adverse event (graded using CTCAE version 5.0), a hospitalization for safety reasons, or death from any cause, whichever occurs first.
Time to clinical deterioration | From randomization, to the date of the first clinical deterioration, up to 24 months
  -Time to clinical deterioration is defined by the time between randomization and deterioration of patient's level of functioning determined by the Eastern Cooperative Oncology Group (ECOG) performance status scale. The ECOG, widely accepted in the community of oncology research to assess how the disease affects the daily living abilities of the patient, is composed of 5 levels from grade 0 (fully active, able to carry on all pre-disease performance without restriction) to grade 5 (dead).
Number of treatment lines | Throughout study completion, up to 24 months
  Number of successive treatment lines offered to the patient from randomization to the end of the study.
Incidence of Adverse Events | Throughout study completion, up to 24 months
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline then every 3 weeks, up to 24 months
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life Questionnaire - Breast cancer module (QLQ-BR45) | At baseline then every 3 weeks, up to 24 months
  This EORTC breast cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BR45 incorporates nine multi-item scales to assess body image, sexual functioning, breast satisfaction, systemic therapy side effects, arm symptoms, breast symptoms, endocrine therapy symptoms, skin mucosis symptoms, endocrine sexual symptoms. In addition, single items assess sexual enjoyment, future perspective and being upset by hair loss. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. Higher scores indicate more severe symptoms or problems for all items.
Treatment compliance and extent of exposure | Throughout study completion, up to 24 months
  The treatment compliance and extent of exposure will be assess using dose intensity, treatment delays and dose reductions.
Compliance with the use of Cureety digital telemonitoring | Throughout study completion, up to 24 months
  Compliance is measured by the frequency of patient responses to the Cureety telemonitoring questionnaires.
Satisfaction with Cureety telemonitoring | 3 months after randomisation for the patients and 1 year after the site activation for medical team
  Satisfaction with Cureety telemonitoring is measured by the percentage of participants (patients and medical team [including nurse, clinical research associate, and investigators]) satisfied by the regular usage of the Cureety telemonitoring tool.
Patient's global satisfaction with care using the data of the EORTC OUT-PATSAT-35 | 6 months after randomisation
  The OUT-PATSAT35 is a 35-item satisfaction with care questionnaire measuring cancer outpatients' perception of hospital doctors and nurses, as well as aspects of care organisation and services. Each item is rated from 1 to 5 (bad to excellent).
Socio-economic impact of digital telemonitoring | Throughout study completion, up to 24 months after randomization
  Socio-economic impact of digital telemonitoring will be assessed using the number of days of hospitalization and the number of unscheduled hospitalizations and emergency consultations

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme MARTIN-BABAU, MD, Principal Investigator — Armorican Centre for Radiotherapy, Medical Imaging and Oncology, CARIO, Plérin; Florence JOLY, MD, Principal Investigator — François Baclesse Center, Caen; Frédéric FITENI, MD, Principal Investigator — University hospital of Nîmes
Locations (51):
- France (51):
  - Institut de Cancérologie des Hauts-de-France (ICHF), Arras
  - Centre Hospitalier d'Auxerre, Auxerre
  - Sainte Catherine - Institut du Cancer Avignon Provence, Avignon
  - CH Aunay-Bayeux, Bayeux
  - Centre Hospitalier Simone Veil de Beauvais, Beauvais
  - ICHF - Centre Pierre Curie, Beuvry
  - Hôpital Simone Veil de Blois, Blois
  - Polyclinique bordeaux nord, Bordeaux
  - Centre Hospitalier Fleyriat, Bourg-en-Bresse
  - Centre de Cancérologie Privé de Caen Maurice Tubiana, Caen
  - Centre Francois Baclesse, Caen
  - Centre hospitalier de Carcasonne, Carcassonne
  - Recherche Oncologie Clinqiue 37 (ROC 37), Chambray-lès-Tours
  - CH de Cholet, Cholet
  - CH Colmar, Colmar
  - Groupe Hospitalier Public du Sud de l'Oise (GHPSO), Creil
  - Centre Georges François Leclerc, Dijon
  - Institut Andrée Dutreix, Dunkirk
  - CH Annecy Genevois, Épagny
  - Centre Hospitalier Intercommunal de Fréjus Saint Raphael, Fréjus
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - CHU de la réunion, La Réunion
  - Clinique Sainte Clotilde, La Réunion
  - Groupe Hospitalier de La Rochelle-Ré-Aunis, La Rochelle
  - CHU Grenoble Alpes, La Tronche
  - Centre Hospitalier Louis Pasteur, Le Coudray
  - Centre Hospitalier Le Mans, Le Mans
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - GHBS Lorient, Lorient
  - Centre Leon Berard, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHI de Mont-de-Marsan et du Pays des Sources, Mont-de-Marsan
  - Centre de Cancérologie du Grand Montpellier, Montpellier
  - Hôpital Privé du Confluent, Nantes
  - Clinique Ambroise-Pare Hartmann, Neuilly-sur-Seine
  - Hôpital Américain de PARIS, Neuilly-sur-Seine
  - CHU de Nimes, Nîmes
  - CHR Orleans, Orléans
  - CHP Sainte-Marie, Osny
  - Diaconesses Croix Saint-Simon Hospital Complex, Paris
  - Centre hospitalier de Pau, Pau
  - CARIO - Hopital Privé des Cotes d'Armor, Plérin
  - CHU de Poitiers, Poitiers
  - Institut Godinot, Reims
  - Clinique Mathilde - Les Hôpitaux Privés Rouennais, Rouen
  - CHU de Saint-Etienne, Saint-Etienne
  - Hia Begin, Saint-Mandé
  - CHU de Tours, Tours
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.